CLINICAL TRIAL: NCT00289666
Title: A Prospective Study to Determine the Effect of Positive Airway Pressure on Heart Rate Variability in Individuals With Obstructive Sleep Apnea
Brief Title: The Effect of Positive Airway Pressure on Heart Rate Variability
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Raelene Maser, Associate Professor, Christiana Care Health Services
Other Study IDs: 23011
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2008-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Disorder; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to determine the effect of continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BiPAP) on heart rate variability (HRV) in patients with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Visit 1: You will come to the Diabetes and Metabolic Research Center having refrained from taking your routine medications and having not eaten in the last 8 hours, avoided using caffeine-containing beverages and tobacco products in the last 10 hours, and having had no alcoholic beverages in the last 24 hours. In addition, you should refrain from taking any nonprescription drugs and avoid engaging in any vigorous exercise for 48 hours before testing.

For those individuals who have diabetes, a letter or direct verbal permission will be obtained, prior to coming to this study visit, from your eye doctor indicating that you can take part in one of the tests listed below. During this visit, an electrocardiogram (EKG, usual heart rhythm test performed in a doctor's office) will be performed. Your heart rate will also be measured for six minutes with an EKG machine while breathing as deeply as possible. This test, which will be performed twice, will tell whether or not the nerves that go to the heart are normal. You will be asked to blow into a plastic tube for 15 seconds (this is the test for which we will obtain the eye doctor's permission for individuals with diabetes). Your heart rate will be measured during and for 60 seconds after you have finished blowing. This test, which will be performed twice, will tell if the nerves that go to blood vessels are normal. Your blood pressure will be measured four times, one minute apart, while you are lying down. You will then be asked to stand up and your blood pressure will again be measured four more times, each time one minute apart. Change in your heart rate will also be determined as you go from lying down to standing. All individuals will have a fingerstick blood sugar level performed prior to the performance of the tests describe above.

You will have about 2 tablespoons of blood drawn. This blood will be stored (frozen) in case possible risk factors of reduced heart rate variability are discovered in the future. A random urine sample will be stored (frozen) for potential examination for microalbuminuria (protein in the urine) or other possible risk factors. At this visit, we will give you a container with instructions for collecting urine for 24-hours. You will also be given some dietary suggestions (e.g., eating a liberal salt diet) that we would like you to follow for 3-days prior to the 24-hour collection of urine. For individuals with diabetes, a small portion of blood will be checked to determine your blood sugar control level.

Standard medical history questions will be asked during this visit along with questions that assess the likelihood of you falling asleep in various situations. Your medical records from your pulmonary doctor will be reviewed for information about the results of the sleep study you had that determined you have a sleep disorder. You will be asked to keep a diary everyday, for the first six weeks, of how many hours per night you use the treatment for your sleep disorder. This visit will last approximately 1-1 ½ hours.

Visit 2: Within 1-48 hours of completion of the 24-hour urine collection and before you begin treatment for your sleep disorder, you will need to bring the urine specimen to the Diabetes and Metabolic Research Center. A part of this urine will be stored (frozen) for possible testing of a hormone called aldosterone, substances filtered by the kidneys (salt and creatinine), and other potential risk factors. Also at this visit, about 2 tablespoons of blood will be drawn and stored for potential testing of a protein in the blood called renin. You should continue the dietary suggestions (e.g., liberal salt diet) given for the collection of the 24-hour urine until the blood is collected. A part of the blood drawn during this visit will also be stored (frozen) in case potential risk factors of heart rate variability are discovered in the future. This visit will last approximately 15 minutes.

Since some drugs can affect how much your heart speeds up and slows down, if your doctor adds a new drug or changes the dosage of any current drugs you may not be able to continue in this study. Please inform a member of the research staff when your doctor makes any change in your medications.

Before coming to the Diabetes and Metabolic Research Center for visit 3, we will need to determine if you have used your device for the treatment of your sleep disorder enough during the six week period. Therefore, a member of the research staff will call you on a weekly basis to ask you to tell us the information that you have recorded in your diary with regard to how often you used the device for the treatment of your sleep disorder.

Visit 3 (approximately six weeks after you begin treatment for your sleep disorder): If you have used the device that is being used to treat your sleep disorder enough, you will be invited to come for visit 3. All of the tests performed during the first visit will be performed again during visit 3. Thus, you will need to follow the same instructions about food, medicine, and exercise as described under visit 1 before coming to visit 3. You will again have a fingerstick blood sugar level performed. In addition, about 2 tablespoons of blood will be drawn. This blood and a random urine sample will be stored (frozen) in case possible risk factors of reduced heart rate variability are discovered in the future and in case these factors need to be examined before and after treatment for a sleep disorder. The same questions asked with regard to the likelihood of you falling asleep in various situations will be asked. This visit will last approximately 1-1 ½ hours.

Visit 4 (approximately 18-months after you begin treatment for your sleep disorder): If you continue to use the device that is being used to treat your sleep disorder for 18-months, you will be invited to come for visit 4. All of the tests performed during the first visit will be performed again during visit 4. Thus, you will need to follow the same instructions about food, medicine, and exercise as described under visit 1 before coming to visit 4. You will again have a fingerstick blood sugar level performed. In addition, about 2 tablespoons of blood will be drawn. This blood and a random urine sample will be stored (frozen) in case possible risk factors of reduced heart rate variability are discovered in the future and in case these factors need to be examined before and after treatment for a sleep disorder. For individuals with diabetes, a small portion of blood will be checked to determine your blood sugar control level. The same questions asked with regard to the likelihood of you falling asleep in various situations will be asked again. This visit will last approximately 1-1 ½ hours.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-75 years old.
* Individuals with diagnosed OSA.

Exclusion Criteria:

* 1. Individuals who are receiving treatment for OSA, excluding those being treated by weight loss.

  2. Individuals who have had pharyngeal surgery (i.e., uvulopalatopharyngoplasty).

  3. Individuals who have arterial oxygen desaturation episodes or apneic episodes not felt to be due to OSA.

  4. Individuals whose treatment dosage changes 2 months prior to, or during, the study for antihypertensive and antidiabetic medications and the following medications that may affect the autonomic nervous system: anti-tuberculosis drugs, nitrofurantoin, metronidazole, chloramphenicol, perhexiline maleate, cordarone, clofibrate, tricyclic antidepressants, phenytoin, barbiturates, neuroleptic drugs, antiparkinsonism drugs, and nitrated drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Care
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-03 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raelene E Maser, PhD, Principal Investigator — University of Delaware
Locations (1):
- Christiana Care Health Service, Newark, Delaware, United States

REFERENCES:
- [Result] Maser RE, Lenhard MJ, Rizzo AA, Vasile AA. Continuous positive airway pressure therapy improves cardiovascular autonomic function for persons with sleep-disordered breathing. Chest. 2008 Jan;133(1):86-91. doi: 10.1378/chest.07-1580. Epub 2007 Oct 20. PMID 17951618